CLINICAL TRIAL: NCT06565884
Title: A Prospective, Randomized, Rate-blind, Multicenter, Optimity-designed Clinical Trial Evaluating the Safety and Efficacy of RFskin Therapy Devices for the Reduction of Skin Wrinkles
Brief Title: Study on the Safety, Efficacy of Home RF Cosmetic Instrument in the Treatment of Facial or Periorbital Wrinkles（F-MFR300-RD-003）
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flossom (GD) Beauty Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F-MFR300-RD-003
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Skin Wrinkles
Keywords: Rf beauty device for home use; Treatment of facial or periorbital wrinkles

STUDY DESIGN:
Intervention Model Description: The method of randomized control and evaluator blindness is suitable for screening A total of 224 subjects were enrolled and randomly divided into control group and experiment according to 1:1 ratio Group)
Who Masked: Outcomes Assessor
Masking Description: Three doctors set up a blind evaluation group to evaluate the photos of the subjects before and after receiving the device treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home radiofrequency skin treatment instrument (Experimental): Radiofrequency skin therapy instrument with medical ultrasound coupler is used for 20 minutes a day, 5 days a week
  Interventions: Device: Home radiofrequency skin treatment instrument
- Medical ultrasound coupler (Placebo Comparator): Medical ultrasound coupler is applied to the face for 20 minutes a day, 5 days a week
  Interventions: Other: Ultrasonic coupler for medical purposes

INTERVENTIONS:
Device: Home radiofrequency skin treatment instrument — Subjects in the experimental group were treated with the test instrument combined with medical ultrasonic coupler for 5 days a week according to the prescribed use method (duration of use: 10 minutes for the whole face, continuous use twice a day, a total of 20 minutes) for 12 weeks. To evaluate the reduction of wrinkles before and after treatment and the changes of laboratory instruments.
  Arms: Home radiofrequency skin treatment instrument
Other: Ultrasonic coupler for medical purposes — In control group, medical ultrasonic coupler was evenly applied on face and orbit for 5 days a week (duration: 20 minutes) for 12 consecutive days Week. To evaluate the reduction of wrinkles and the change of laboratory instruments before and after use.
  Arms: Medical ultrasound coupler

SUMMARY:
This is a multicenter trial with randomized control and evaluator blind method, which meets the screening criteria total of 224 subjects were enrolled and randomly divided into control group and experiment according to 1:1 ratio Group), the subjects in the control group used medical ultrasonic coupler, and the subjects in the test group used test instruments Combined with medical ultrasonic coupler, use 5 days per week according to the prescribed use method (duration:Use the whole face for 10 minutes, use twice a day, a total of 20 minutes), continuous use 12Week. The changes of relevant clinical indicators and laboratory instrument measurements were evaluated.

Objective : To evaluate the efficacy of radiofRF in reducing skin wrinkles and treating loose skin after 12 weeks of use of the test product Effectiveness and safety of relaxation and firming of skin tissue.

The subjects were adults aged 18 years and above, regardless of gender, and had obvious wrinkles on the skin around the face and eyes (according to the selection Standard confirmation).

DETAILED DESCRIPTION:
The purpose of the clinical trial was to see if home radiofrequency beauty devices were effective in treating adults for reducing skin wrinkles. It will also learn about the safety of home RF beauty devices. The main questions it aims to answer are:

1. Reduction of facial or periocular wrinkles based on Fitzpatrick score (12 weeks);
2. Possible adverse reactions and satisfaction survey during the use of subjects; The researchers will compare the radiofrequency beauty device group with the control group (only medical ultrasonic coupling) to verify whether the home radiofrequency beauty device is effective in reducing skin wrinkles.

Participants will:

Receive home treatment according to the experimental group and continue to use it for 12 weeks.

At the 6th and 12th week, they will visit the medical institution for questionnaire survey and skin test.

Keep a diary of their symptoms and the number of times they use radiofrequency beauty device or medical ultrasonic coupling.

ELIGIBILITY:
Inclusion Criteria:

* (1) Adults aged 18 and above, male or female;
* (2) Fitzpatrick's wrinkles and elasticity scores around the face and eyes were 2-7 points (on-site assessment);
* (3) To avoid sun exposure during the test;
* (4) Be able to read Chinese and accurately understand, and sign the informed consent of the test;
* (5) can cooperate with and participate in the test return visit time, and timely reflect their own health status or any changes in drugs, adverse reaction symptoms;
* (6) Urine pregnancy reaction is negative (women of childbearing age).

Exclusion Criteria:

* (1) Abnormal vital signs (blood pressure, pulse, body temperature), except for minor abnormalities that are not clinically significant as determined by the doctor;
* (2) There is a pacemaker or internal defibrillator in the body, or any other active electrical implant anywhere in the body;
* (3) The treatment area has permanent implants, such as metal plates and screws (e.g. dentures, metal teeth), silicone implants or injected chemicals;
* (4) There is or has been a history of skin cancer, or any other type of cancer, or malignant pre-nevus;
* (5) serious comorbidities, such as heart disease, epilepsy, high blood pressure and liver or kidney disease;
* (6) Plan to become pregnant or breastfeed during the study period, or less than 6 months after delivery;
* (7) Have a history of bleeding and clotting, or long-term use of anticoagulation and antiplatelet drugs (aspirin ≤81mg daily is not excluded);
* (8) Suffering from autoimmune diseases;
* (9) have an immunosuppressive disease such as AIDS, or an impaired immune system caused by the use of immunosuppressive drugs (investigators' judgment);
* (10) Subjects with a history of heat-stimulated disease, such as recurrent herpes simplex in the treatment area, should only be treated after a preprevention regimen;
* (11) Poor control of diseases related to the endocrine system as determined by the investigator, such as diabetes or thyroid dysfunction;
* (12) Any active condition in the treatment area identified by the investigator, such as ulcers, eczema, or other skin lesions;
* (13) A history of skin diseases, such as keloid, abnormal wound healing, psoriasis, etc.;
* (14) Any invasive or non-invasive treatment (such as hair removal, light rejuvenation, microneedles or chemical exfoliation, etc.) in the treated area within 3 months prior to treatment;
* (15) Received RF microneedle therapy, injection of fillers or botulinum toxin within 6 months prior to treatment;
* (16) Receive semi-permanent fillers (poly-l-lactic acid, calci-hydroxyphospholite, etc.) within 24 months before treatment;
* (17) Have undergone facial medical or cosmetic surgery (e.g. eyelid/ eyebrow surgery, periorbital or perioral soft tissue enhancement, permanent fillers, permanent makeup, tattoos, etc.);
* (18) Use of drugs that may trigger photosensitization during the study period (such as quinolones, aspirin, hyd rochlorothiazide or furosemide);
* (19) Use of any medications that affect skin characteristics (e.g., vitamin A, steroids, thyroid medications, etc.) in the past 6 months;
* (20) Participate in a clinical trial of another drug or device in which the last treatment of the investigational drug/device occurred 3 months before the start of treatment in the study;
* (21) Plan to change previously used skin care products during the study period;
* (22) Other conditions deemed unsuitable for inclusion by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Wrinkle reduction efficiency based on Fitzpatrick score | 12th week
  After 12 weeks of treatment, wrinkles were more severe on a 0-9 scale (Fitzpatrick scale) Percentage of subjects with at least one grade (1 point) reduction at baseline.

SECONDARY OUTCOMES:
Wrinkle reduction efficiency based on Fitzpatrick score | 6th week
  After 6 weeks of treatment, wrinkles were more severe on a 0-9 scale (Fitzpatrick scale) Percentage of subjects with at least one grade (1 point) reduction at baseline.
R2 values measured by the Cutometer dual MPA580 | 6th week\12th week
  The R2 values of the two groups were compared after 6 weeks /12 weeks after using the RF instrument.
F4 values measured by the Cutometer dual MPA580 | 6th week\12th week
  The F4 values of the two groups were compared after 6 weeks /12 weeks after using the RF instrument.
PRIMOS-CR measures the length of skin wrinkles | 6th week\12th week
  PRIMOS-CR measured crow's feet and compared the number of wrinkles between the two groups Quantity
PRIMOS-CR measures the length and number of skin wrinkles | 6th week\12th week
  PRIMOS-CR measured under-eye lines and compared the number of wrinkles between the two groups Quantity
PRIMOS-CR measures the length and number of skin wrinkles | 6th week\12th week
  PRIMOS-CR measured crow's feet and compared the number of wrinkles between the two groups length
PRIMOS-CR measures the length and number of skin wrinkles | 6th week\12th week
  PRIMOS-CR measured under-eye lines and compared the number of wrinkles between the two groups length
Lower face sag evaluation | 6th week\12th week
  According to the researchers' Skin Aging Atlas (R.Busin, F.folament), skin aging Tu Volume 2 Asian Edition). Translated by Qiu Huixia et al. [M]. Paris: MED 'com, 2010.) " To assess the severity of the subject's lower bilateral sagging.
Subject satisfaction evaluation | 6th week\12th week
  The participants received a questionnaire at the last visit, which mainly included the skin improvement effect of the product And the satisfaction degree of ease of operation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lai, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No